CLINICAL TRIAL: NCT07333924
Title: How Can we Best Communicate the Findings of Systematic Reviews to the Public? A Study Within A Review
Brief Title: Randomised Study Within a Review (SWAR) to Compare Communication of the Findings of Systematic Reviews to the Public by Plain Language Summary or Video Abstract
Acronym: SWAR02-2026
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Aberdeen Belfast Evidence Collaboration (Unknown)
Responsible Party: Principal Investigator, Mike Clarke, Chair, Research Methodology, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SWAR02-2026
Record Dates: First submitted 2025-12-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Behavioral Changes
Keywords: Plain language summary; Animated video; Study Within a Review (SWAR); Systematic reviews; Evidence synthesis; Public understanding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reading group (Active Comparator): Written summary of a systematic review
  Interventions: Other: Plain language summary
- Video group (Experimental): Video summary of a systematic review
  Interventions: Other: Animated video

INTERVENTIONS:
Other: Plain language summary — A written summary of the systematic review.
  Arms: Reading group
Other: Animated video — An animated video summary of the systematic review.
  Arms: Video group

SUMMARY:
A systematic review is a type of research that collects and analyses all the existing studies on a specific topic in a structured and organised way. Instead of just looking at one study, it combines results from many studies to get a clearer, more reliable answer to a question. However, the complex language used in systematic reviews often makes them inaccessible to the public, highlighting the need for effective communication strategies, particularly for reviews relating to health and social care or public health. However, there is limited research exploring alternative ways to present research articles, with only a few delivery methods studied so far. It remains unclear how different styles of communicating might effectively convey scientific findings accurately or enhance public engagement and understanding of complex topics.

Studies Within A Review (SWARs) are studies which are embedded into a systematic review and aim to form an evidence base to improve how we plan, do, and share systematic reviews. SWARs offer a promising way of improving the methodology of systematic reviews and dissemination of their findings.

This randomised trial aims to address the current research gap by identifying the effectiveness of two different ways to communicate systematic review findings to the public and determining which methods are more suitable for different audiences: participants will be asked to read a summary or watch an animated video of a summary of both reviews and then complete a questionnaire about the reviews' findings and conclusions. The study will assess outcomes such as comprehension, perceived understanding, engagement, and interest of participants in reading the full reviews.

By evaluating the impact of different communication strategies, this study aims to strengthen the evidence base for methods to communicate complex scientific findings to the public. The results are expected to provide valuable insights for optimising the communication of the key findings of systematic reviews, ensuring that summaries are clear, engaging and accessible.

DETAILED DESCRIPTION:
This randomised Study Within a Review (SWAR) will address the uncertainty in communicating the findings of systematic reviews by comparing the effectiveness of two communication methods. We will evaluate participants' understanding of the key findings from two systematic reviews and their interest in seeking further information. These systematic reviews (summarised below), while covering entirely different topics, are both complex and highly relevant to public health.

Systematic Review 1: Clinical Utility of Biomarkers for Outcomes Prediction in Adults with Suspected Sepsis Presenting to the Emergency Department Sepsis is associated with a high mortality rate, and early detection and diagnosis is crucial. This review aimed to determine whether biomarkers measured in patients presenting to an emergency department with suspected sepsis may predict deterioration, including mortality, critical care admission, organ failure, and septic shock.

Systematic Review 2: Local antibiotics for patients undergoing surgery for open fractures Open fractures are serious injuries where the bone breaks through the skin, often leading to complications like infection. Treating these injuries can be complex and expensive, with many patients needing multiple operations and ongoing care. This review sought to determine if there is evidence that local antibiotics may reduce infection in people who are having surgery for open fractures.

The objectives of this study are

1. To determine whether a plain language summary or animated video summary is more effective in conveying the core message of a systematic review.
2. To compare the effects of the two methods on perceived understanding, engagement, and interest in reading the full text of the systematic review

Recruitment plan We will recruit using multiple methods. The study will be advertised through various channels, including posters displayed in common areas of the host university (Queen's University Belfast) and other popular locations across Belfast, social media platforms such as Instagram, Twitter and LinkedIN, and word of mouth. People interested in taking part will be able to contact the research team directly using the provided contact details.

Study procedures Potential participants will email or click on a QR code on the study posters (in person or via social media), which will bring them to the study information and a consent form. They will read that their participation will take a maximum of 30 minutes for the first round, and that they will asked to participate in a second round of questions 1 to 2 weeks later, which can be done via telephone pr email if preferred and would take less than 10 minutes. They will be asked to include their first name or a nick-name and contact details (email or telephone) so that the research team can contact them. Participants will also be asked to answer some additional questions to collect their age, scientific education and whether they had any scientific training after secondary education, and if they feel they know anything about the review topics.

The research team will contact those who have volunteered and have agreed to participate by email or telephone. A meeting will be arranged for a public space where they can sit comfortably with minimal noise and distractions. Participants will be randomly assigned to one of two groups: either the Reading Group or the Video Group (as shown in Table 1). Within each group, participants will be randomly assigned to start with Review 1 or Review 2. Once people are enrolled in the study, they will be assigned a unique ID number.

The intervention will be administered on a tablet computer. Those in the Reading Group will read the summary of their first review on the tablet and then answer related questions. After completing this review, they will read the summary of their second review and answer corresponding questions. Participants in the Video Group will use headphones while watching the Animated Video summary of their first review and then answer related questions on the tablet. After completing that review, they will watch an Animated Video summary of their second review and answer corresponding questions.

Participants will be reminded that they will be contacted for a follow-up assessment 1-2 weeks after the initial session. They will be contacted using the contact method they provided during the consent process. Follow-up can be face-to-face, or by email or phone.

Statistical analysis Participants' responses related to the Plain Language Summary and Animated Video Summary of Review 1 and Review 2 will be compared. Differences between groups will be assessed using the T-test/Mann-Whitney U test (as appropriate). A convenience sample of 100 participants will be sought, based on the time available for the researcher to conduct the data gathering.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years+)
* Any gender
* Able to read and understand English
* Willing to read and listen to review summaries, and answer questions
* Provide informed consent to participate

Exclusion Criteria:

* People with learning difficulty
* People who do not read or understand English
* People with hearing or visual impairment
* People under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Immediate comprehension of the information presented in the review summary. | Immediately after interaction with the summary.
  A multiple-choice question is included to assess participants' understanding of the primary focus of the research by asking them to choose from a list of topics about the focus of the review, only one of which is correct. There are also five questions presented as statements relating to specific content from the review summary and participants are required to indicate whether each statement is true or false. The unit of measure will be the proportion of participants who select the correct answer to each question. The assessment tool was adapted from Bredbenner K, Simon SM. Video abstracts and plain language summaries are more effective than graphical abstracts and published abstracts. PloS ONE 2019;14(11):e0224697.
Retention of the participant's comprehension of the information presented in the review summary | 1 to 2 weeks after interaction with the summary.
  Participants will answer the same six questions that were used to assess their comprehension immediately after their interaction with the summary. This will include a multiple-choice question asking them to choose from a list of topics about the focus of the review, only one of which is correct. There are also five questions presented as statements relating to specific content from the review summary and participants are required to indicate whether each statement is true or false. The unit of measure will be the proportion of participants who select the correct answer to each question. The assessment tool was adapted from Bredbenner K, Simon SM. Video abstracts and plain language summaries are more effective than graphical abstracts and published abstracts. PloS ONE 2019;14(11):e0224697.

SECONDARY OUTCOMES:
Participant's perceived understanding (i.e. how well they believe they understood the review summary) | Immediately after interaction with the summary.
  Participants will be asked to rate their understanding of the review on a 5-point scale: 0 = Not a Bit; 1 = A Bit; 2 = Average; 3 = Mostly; 4 = Very Much.
  The unit of measure will be the mean and median for these scores within each intervention group. The assessment tool was adapted from Bredbenner K, Simon SM. Video abstracts and plain language summaries are more effective than graphical abstracts and published abstracts. PloS ONE 2019;14(11):e0224697.
Participant's enjoyment of their interaction with the summary | Immediately after interaction with the summary.
  Participants will be asked to rate the extent to which they found the review summary engaging on a 5-point scale: 0 = Not a Bit; 1 = A Bit; 2 = Average; 3 = Mostly; 4 = Very Much.
  The unit of measure will be the mean and median for these scores within each intervention group. The assessment tool was adapted from Bredbenner K, Simon SM. Video abstracts and plain language summaries are more effective than graphical abstracts and published abstracts. PloS ONE 2019;14(11):e0224697.
Participant's interest in reading the full text of the systematic review after their interaction with its summary | Immediately after interaction with the summary.
  Participants will be asked to rate their interest in finding out more about the systematic review on a 5-point scale: 0 = Not a Bit; 1 = A Bit; 2 = Average; 3 = Mostly; 4 = Very Much.
  The unit of measure will be the mean and median for these scores within each intervention group. The assessment tool was adapted from Bredbenner K, Simon SM. Video abstracts and plain language summaries are more effective than graphical abstracts and published abstracts. PloS ONE 2019;14(11):e0224697.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maguire LK, Clarke M. How much do you need: a randomised experiment of whether readers can understand the key messages from summaries of Cochrane Reviews without reading the full review. J R Soc Med. 2014 Nov;107(11):444-9. doi: 10.1177/0141076814546710. Epub 2014 Oct 23. PMID 25341445
- [Background] Devane D, Burke NN, Treweek S, Clarke M, Thomas J, Booth A, Tricco AC, Saif-Ur-Rahman KM. Study within a review (SWAR). J Evid Based Med. 2022 Dec;15(4):328-332. doi: 10.1111/jebm.12505. Epub 2022 Dec 13. No abstract available. PMID 36513956
- See also: SWAR02 original outline — https://www.qub.ac.uk/sites/TheNorthernIrelandNetworkforTrialsMethodologyResearch/FileStore/SWARFileStore/Filetoupload695595en.pdf